CLINICAL TRIAL: NCT02985346
Title: Sun Yat-sen Memorial Hospital
Brief Title: Efficacy of Bone Marrow Mesenchymal Stem Cell in Pulmonary Hemosiderosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weiping Tan, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTan
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Idiopathic Pulmonary Hemosiderosis
Keywords: Idiopathic pulmonary hemosiderosis; Bone marrow mesenchymal stem cells
MeSH Terms: conditions — Hemosiderosis, Pulmonary

ARMS (2):
- BMSC group (Experimental): Patients received Bone marrow mesenchymal stem cells (BMSC) plus standard treatment
  Interventions: Biological: Bone marrow mesenchymal stem cells in treatment of Idiopathic pulmonary hemosiderosis
- Control group (Active Comparator): Patients received standard treatment
  Interventions: Biological: Bone marrow mesenchymal stem cells in treatment of Idiopathic pulmonary hemosiderosis

INTERVENTIONS:
Biological: Bone marrow mesenchymal stem cells in treatment of Idiopathic pulmonary hemosiderosis

SUMMARY:
Pulmonary hemosiderosis (PH) is a pulmonary hemosiderin deposition which caused by alveolar capillary hemorrhage. PH is easy to recurrent and can lead to pulmonary fibrosis and insufficiency if the disease was poor controlled. Steroid is the most common drug that was administered in acute phase of the disease. However, considered the side-effects, steroid is not suitable for long-time maintenance. Therefore, it is necessary to explore a new therapy. Bone marrow mesenchymal stem cells (BMSC) are a kind of adult stem cells with high self-renewal and multi-directional differentiation potential in bone marrow. It has become a hot topic in immunosuppressive and tissue repair therapy in recent years. To date, homing, colonization and differentiation of BMSCs in the lung have been observed in animal models of pulmonary hypertension, radiation pneumonitis and pulmonary fibrosis. It had been reported that BMSC transplantation in acute lung injury in mice, inflammation of lung injury can significantly improve. The aim of this study is to explore the effect of BMSC on PH and its mechanism, and to explore a new way to promote the repair of IPH. It is expected to improve the status of IPH therapy in children, especially improve the prognosis of refractory PH.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Pulmonary hemosiderosis at an age less than 18 years.

Exclusion Criteria:

* Patients who cannot finish the established causes or die during the causes.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 3-6 months

REFERENCES:
- [Background] Byrd RB, Gracey DR. Immunosuppressive treatment of idiopathic pulmonary hemosiderosis. JAMA. 1973 Oct 22;226(4):458-9. No abstract available. PMID 4800237
- [Background] Airaghi L, Ciceri L, Giannini S, Ferrero S, Meroni PL, Tedeschi A. Idiopathic pulmonary hemosiderosis in an adult. Favourable response to azathioprine. Monaldi Arch Chest Dis. 2001 Jun;56(3):211-3. PMID 11665500
- [Background] Calabrese F, Giacometti C, Rea F, Loy M, Sartori F, Di Vittorio G, Abudureheman A, Thiene G, Valente M. Recurrence of idiopathic pulmonary hemosiderosis in a young adult patient after bilateral single-lung transplantation. Transplantation. 2002 Dec 15;74(11):1643-5. doi: 10.1097/00007890-200212150-00027. PMID 12490803
- [Background] Chen RL, Chuang SS. Silent idiopathic pulmonary hemosiderosis with iron-deficiency anemia but normal serum ferritin. J Pediatr Hematol Oncol. 2007 Jul;29(7):509-11. doi: 10.1097/MPH.0b013e3180950372. No abstract available. PMID 17609633
- [Result] Rojas M, Xu J, Woods CR, Mora AL, Spears W, Roman J, Brigham KL. Bone marrow-derived mesenchymal stem cells in repair of the injured lung. Am J Respir Cell Mol Biol. 2005 Aug;33(2):145-52. doi: 10.1165/rcmb.2004-0330OC. Epub 2005 May 12. PMID 15891110
- [Result] Wang G, Bunnell BA, Painter RG, Quiniones BC, Tom S, Lanson NA Jr, Spees JL, Bertucci D, Peister A, Weiss DJ, Valentine VG, Prockop DJ, Kolls JK. Adult stem cells from bone marrow stroma differentiate into airway epithelial cells: potential therapy for cystic fibrosis. Proc Natl Acad Sci U S A. 2005 Jan 4;102(1):186-91. doi: 10.1073/pnas.0406266102. Epub 2004 Dec 22. PMID 15615854
- [Result] Lee JW, Fang X, Gupta N, Serikov V, Matthay MA. Allogeneic human mesenchymal stem cells for treatment of E. coli endotoxin-induced acute lung injury in the ex vivo perfused human lung. Proc Natl Acad Sci U S A. 2009 Sep 22;106(38):16357-62. doi: 10.1073/pnas.0907996106. Epub 2009 Aug 31. PMID 19721001
- [Result] Knight DA, Rossi FM, Hackett TL. Mesenchymal stem cells for repair of the airway epithelium in asthma. Expert Rev Respir Med. 2010 Dec;4(6):747-58. doi: 10.1586/ers.10.72. PMID 21128750
- [Result] Hoffman AM, Paxson JA, Mazan MR, Davis AM, Tyagi S, Murthy S, Ingenito EP. Lung-derived mesenchymal stromal cell post-transplantation survival, persistence, paracrine expression, and repair of elastase-injured lung. Stem Cells Dev. 2011 Oct;20(10):1779-92. doi: 10.1089/scd.2011.0105. Epub 2011 Jul 6. PMID 21585237
- [Result] Liu AR, Liu L, Chen S, Yang Y, Zhao HJ, Liu L, Guo FM, Lu XM, Qiu HB. Activation of canonical wnt pathway promotes differentiation of mouse bone marrow-derived MSCs into type II alveolar epithelial cells, confers resistance to oxidative stress, and promotes their migration to injured lung tissue in vitro. J Cell Physiol. 2013 Jun;228(6):1270-83. doi: 10.1002/jcp.24282. PMID 23154940